CLINICAL TRIAL: NCT02632682
Title: Real-time Diagnosis of Barrett's Esophagus: Comparing Confocal Laser Endomicroscopy With Conventional Histology for the Identification of Specialized Intestinal Metaplasia
Brief Title: Confocal Laser Endomicroscopy vs Conventional Histology for the Identification of Intestinal Metaplasia
Status: Completed | Type: Observational
Sponsor: Minnesota Institute for Minimally Invasive Surgery (Other)
Collaborators: The Oregon Clinic (Other)
Responsible Party: Sponsor
Other Study IDs: CLE-08
Record Dates: First submitted 2015-12-04; First posted 2015-12-17 (Estimated); Last update posted 2016-12-02 (Estimated); Status verified 2016-11

CONDITIONS: Barrett's Esophagus
Keywords: probe-based confocal laser endomicroscopy
MeSH Terms: conditions — Barrett Esophagus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Real-time Diagnosis of Barrett's Esophagus: Comparing Confocal Laser Endomicroscopy with Conventional Histology for the Identification of Specialized Intestinal Metaplasia

DETAILED DESCRIPTION:
The incidence of esophageal adenocarcinoma has risen over 800% over the past several decades and is associated with a high mortality rate. Barrett's esophagus (BE) has been identified as the number one risk factor for the development of esophageal adenocarcinoma. Gastroesophageal reflux disease (GERD) has been identified as the major risk factor for development of BE. Current guidelines for BE diagnosis and surveillance, according to the Seattle protocol, include four-quadrant random biopsies at 2-cm intervals (1-cm intervals if suspected high grade intraepithelial neoplasia). This random biopsy protocol can be time-consuming, expensive, and prone to sampling error, as very little of the esophageal surface area is actually sampled. Probe-based confocal laser endomicroscopy (pCLE) generates optical biopsies, providing physicians with microscopic images of tissue instantaneously and in a minimally invasive manner. Comparing pCLE with conventional histology for the identification of specialized intestinal metaplasia has the potential to result in a new standard of care for the diagnosis of BE. The aim of this study is to compare pCLE to traditional tissue biopsies for the diagnosis of BE.

A patient with GERD will be scheduled for upper endoscopy as part of routine evaluation. Routine endoscopy will be performed, including white light and narrow band imaging photo documentation. Probe-based confocal laser endomicroscopy will be performed at the gastroesophageal junction. Biopsies of columnar lined esophagus will then be taken in four quadrants starting at the squamocolumnar junction and proceeding in 1 cm segments to the gastroesophageal junction. Optical biopsy images will be reviewed immediately following endoscopy by endoscopist and later reviewed by blinded independent reviewer. Pathology specimens will be reviewed by a pathologist. The results of the optical biopsies obtained with probe-based confocal laser endomicroscopy will be compared with the pathology results.

ELIGIBILITY:
Inclusion Criteria:

* Age >18; Clinical diagnosis of GERD; Undergoing upper endoscopy for reflux evaluation

Exclusion Criteria:

* Age <18, Contraindication to receiving fluorescein, Inability to provide informed consent, History of esophageal ablation

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: * Age >18
  * Clinical diagnosis of GERD
  * Undergoing upper endoscopy for reflux evaluation
Sampling Method: Non-Probability Sample
Enrollment: 172 (Actual)
Dates: Start 2016-02; Primary Completion 2016-08 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Probe-based confocal laser endomicroscopy (pCLE) will be compared to standard histologic analysis in the evaluation of Barrett's esophagus. | 8 months
  Metrics for the study will include "positive" or "negative" for Barrett's esophagus.

IPD SHARING:
Plan to Share IPD: No